CLINICAL TRIAL: NCT01318668
Title: An fMRI-study on the Effects of 3'-Aminomethylnicotine-P. Aeruginosa r-Exoprotein a Conjugate Vaccine (NicVAX®) and Placebo on Central Nervous System Activation and Behaviour Following a Nicotine Challenge
Brief Title: A Fmri Study on the Effects of a Conjugate Vaccine and Placebo on CNS Activation and Behavior Following a Nicotine Challenge
Acronym: EPU057
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Principal Investigator, Vuurman, Dr Eric Vuurman, Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: CCMO31915
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Nicotine Dependency; Smoking
Keywords: fmri smoking vaccination mood
MeSH Terms: conditions — Smoking | interventions — Vaccination; NicVAX

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nicotine vaccination (Experimental): 18 week treatment with Nicvax
  Interventions: Biological: vaccination with Nicvax

INTERVENTIONS:
Biological: vaccination with Nicvax — 5 vaccinations of NicVax 400ug (1 ml) over a 18 week period or matching placebo.
  Other Names: NicVAX is a P. earoginosa r-Exoprotein conjugate vaccine.

SUMMARY:
In this study the effects of a nicotine challenge on brain activity, behavior and mood will be evaluated in two groups of healthy volunteers who have a smoking habbit: The first group will undergo a series of treatments with NicVax, aimed at producing nicotine antibodies in the body and preventing nicotine to enter the brain. The second group will receive a placebo treatment. This pre-treatment (vaccination) will take place over a 18-week period. All participants will then undergo two days of testing. On each day the subjects will perform a number of psychomotor and memory tests after a challenge with nicotine (gum) or placebo(gum). Also brain activity will be studied in an fMRI scanner. We expect to see an effect on brain activation and performance only in the placebo-vaccinated group. The Nicvax vaccinated group should show activation and performance comparable to that after challenge with placebo(gum) as in this group nicotine should not cross the blood brain barrier and enter the brain

DETAILED DESCRIPTION:
Rationale: To develop a more effective treatment for nicotine addiction is a public health priority. In order to do so a better understanding is needed of the mechanisms 1) underlying nicotine addiction and 2) the way treatments alter the way nicotine transiently and permanently alters multiple cognitive and executive functions. Most effects of nicotine on the Central Nervous System (CNS) are directly mediated by nicotine molecules. Treatment with 3'aminomethylnicotine P. aeruginosa r-Exoprotein A Conjugate Vaccine (NicVAX™) stimulates the production of nicotine specific antibodies. These antibodies bind the small nicotine molecules, preventing them to cross the Blood Brain Barrier (BBB) and thus preventing CNS stimulation. A nicotine challenge given after vaccination will show no or diminished direct effects of nicotine on CNS stimulation. The blocking effects of the nicotine specific antibodies will be evaluated on several cognitive tasks and on reactivity to smoking-related cues.

Objective: Main aim; to show that NicVAX attenuates nicotine induced CNS effects on brain activation and cognitive performance relative to placebo. The secondary aim is to evaluate how these changes in CNS stimulation alter subjective measures and the addictive properties of nicotine.

Study design: within-subject cross-over double-blind placebo controlled study. Study population: 48 current smokers, male, age 25-40, at least smoking 10 cigarettes /day the last year, in general good health. Additional criteria; 1) No contra-indications for MRI 2) No history of cognitive deficits or brain trauma 3) No use of psychoactive medication 4) No contra-indications for nicotine gum.

Intervention (if applicable): The group will be randomized in two sub-populations. 1) 28 volunteers will receive five injections of 3'aminomethylnicotine P. aeruginosa r-Exoprotein A Conjugate Vaccine (NicVAX™), 2) 20 smokers will receive five injections placebo. On test days both groups will be given a nicotine challenge; a chewing gum either containing nicotine (2mg) or a placebo.

Main study parameters/endpoints: correlation between nicotine specific antibody and 1) the BOLD response during resting state, during the smoking-cue reactivity paradigm and during task performance; in regions of interest associated with the specific tasks; 2) the number of correct response and the reaction time; 3) correlation between nicotine specific antibody and subjective signs of nicotine addiction, measured with several questionnaires.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: participants will complete a medical screening questionnaire (15-30 min) and will undergo a medical screening (45 min; 2 blood samples, a urine sample and an electrocardiogram). Informed consent will be obtained. All participants will be vaccinated with NicVAX or Placebo 5 times on day 0, 28, 56, 84 and 112 (4 weeks in between each injection) During the training session (Day 0; ±1,5 hour) the inclusion/exclusion criteria and baseline laboratory results will be reviewed to ensure that no changes to the participants health and eligibility status occurred since the Screening Visit. Participants will be randomized and receive either one dose NicVAX 400µ in 1 ml or a placebo intramuscular. The cognitive fMRI task will be trained in a dummy scanner, and questionnaires will be completed. Subsequent vaccinations (days 28, 56, 84 and 112) should be given in the alternating deltoid muscle. Participants will be observed for 60 minutes to monitor possible adverse events. Adverse events, vital signs and concomitant medications will be recorded. During each test session (days 133, 140) participants will complete 5 questionnaires (30 minute total) and will perform several cognitive tasks inside the fMRI scanner (scan session in total ~85 min). The last test session (day 140) three blood samples (5-8 ml each) will be taken for nicotine-specific antibody assessment and to monitor changes. In total the study will take 18 hours to complete. The participants will be paid 10 euro/hr as compensation. The risk of vaccination, fMRI scanning and of administration of nicotine 2mg gum (delivering a dose of approximately 1-1.5 mg nicotine to the bloodstream) is negligible for carefully screened participants. The nicotine specific-antibody vaccine has been clinically tested on several occasions; the safety profile was favourable. Local reactogenicity was generally mild to moderate and subsided spontaneously. Vaccinated subjects with the highest antibody levels (top 30%) smoked less cigarettes per day and reported a higher abstinence rate than placebo subjects, establishing proof-of-concept. The group receiving the vaccine could therefore in theory reduce smoking/exposure to tobacco smoke and have consequential health benefits.

ELIGIBILITY:
Inclusion Criteria:

* Health male right handed volunteers between 25-40 years of age.
* Smoking at least 10 cigarettes per day

Exclusion Criteria:

* Contra indications for MRI scanner
* History of neurological or psychiatric disease
* known immunodeficiency
* current use of psychoactive medication
* excessive alcohol use

Ages: 25 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
FMRI | at 18 and 20 weeks post vaccination
  Regional blood oxygenated level dependent (BOLD) response (method: BOLD functional MRI) during resting state and during task performance, in regions of interest, before and after nicotine administration.
Reaction time | at 18 and 20 weeks post vaccination
  Task performance; the number of correct response and the reaction time in a battery of psycho-motor tests.

SECONDARY OUTCOMES:
Mood | 18 and 20 weeks post vaccination
  Mood will be evaluated by means of questionnaires prior to and following the nicotine/placebo challenge

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Havermans A, Vuurman EF, van den Hurk J, Hoogsteder P, van Schayck OC. Treatment with a nicotine vaccine does not lead to changes in brain activity during smoking cue exposure or a working memory task. Addiction. 2014 Aug;109(8):1260-7. doi: 10.1111/add.12577. Epub 2014 Jun 3. PMID 24894701